CLINICAL TRIAL: NCT06217328
Title: A Prospective Randomized Control Trial to Compare the Efficacy of the Revi System Therapy on Versus Off in Relieving Urinary Urge Incontinence Episodes.
Brief Title: RESTORE: An RCT to Evaluate the Efficacy of the Revi System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BlueWind Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G02-CLP-0019
Record Dates: First submitted 2024-01-03; First posted 2024-01-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Urinary Urge Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: All subjects will be implanted with the device and randomized (2:1) to ON vs OFF. After the subjects complete the OFF period, their system will be activated and they will crossover to the ON group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Device: Revi System Treatment Arm (Other): Subjects will be implanted with a Revi System and activation of therapy will occur ~4 weeks post implantation and continue for the duration of the study.
  Interventions: Device: Revi System Treatment
- Device: Revi System - Delayed Activation Control Arm (Other): Subjects will be implanted with a Revi System and activation of therapy will be delayed until 4 months post implantation. At this time the Revi System will be activated to begin therapy and will continue for the duration of the study.
  Interventions: Device: Revi System - Delayed Activation

INTERVENTIONS:
Device: Revi System Treatment — The Revi System is an implantable neuromodulation device placed in the ankle region that is activated by a battery-operated rechargeable external wearable
  Arms: Device: Revi System Treatment Arm
Device: Revi System - Delayed Activation — The Revi System is an implantable neuromodulation device placed in the ankle region that is activated by a battery-operated rechargeable external wearable. The system will be implanted but it will not be turned on until 4 months post implant procedure.
  Arms: Device: Revi System - Delayed Activation Control Arm

SUMMARY:
The Revi System is indicated for the treatment of patients with symptoms of urgency incontinence alone or in combination with urinary urgency.

DETAILED DESCRIPTION:
Prospective, multi-center, open label, post market, randomized controlled trial

To demonstrate superiority of Revi System therapy vs. non active therapy in the treatment of UUI

Treatment Arm:

Device: Revi System Subjects will be implanted with a Revi System and activation of therapy will occur ~4 weeks post implantation and continue for the duration of the study.

Control Arm:

Device: Revi System - Delayed Activation Subjects will be implanted with a Revi System and activation of therapy will be delayed until 4 months post implantation. At this time the Revi System will be activated to begin therapy and will continue for the duration of the study.

Randomization in a 1:2 ratio into either the "control group" or the "treatment group" will be performed in blocks of 3 or 6 randomly, across the study population by a central randomization system. Randomization will be stratified by investigational site.

The study will consist of the following activities:

Visit 1 - Screening

* Potential subjects with UUI, who fulfil basic criteria will be informed of the study and will be invited to sign an informed consent form.
* Demographic information (age, race, height and weight, leg circumference), medical and surgical history and concomitant medication information will be collected.
* Study candidates will be asked to fill out various questionnaires
* Patients will be asked to complete a 3- consecutive day voiding diary.
* Urine sample will be collected, blood will be drawn and a full physical examination, including a PVR measurement and uroflow (in men), will be performed.

Visit 2 - Randomization & Implantation

* 5 ± 4 weeks after starting the diary, eligible subjects will be randomized to either the Treatment or Control (delayed activation) arms (2:1) and will undergo unilateral implantation with the BlueWind Revi System
* Collection of AE and concomitant medication will be performed

Treatment Arm:

Visit 3 - Activation

* After a recovery period of 4-weeks post implantation, subjects will attend the clinic to undergo physical examination and surgical wound check-up.
* Subjects will undergo parameter setting according to the individual patient sensations and will be trained on the use of the system.

Visits 4-11 - Treatment optimization and follow up

* Follow-up visits will be performed at 1, 2, 3, 6, 9, 12, and 24 months post system activation.
* A call visit will be performed at 18-months.
* All follow-up visits will require completion of a 3-day voiding diary by the patient before coming to the visit.
* During each clinic visit, stimulation parameters and level of treatment will be checked and adjusted as needed.

Control Arm:

• After a recovery period of 1-month post implantation, subjects will attend the clinic to undergo physical examination and surgical wound check-up.

Visit 4 - Activation

* After a recovery period of 4-weeks post implantation, subjects will attend the clinic to undergo physical examination and surgical wound check-up.
* Subjects will undergo parameter setting according to the individual patient sensations and will be trained on the use of the system.

Visits 5-12 - Treatment optimization and follow up

* Follow-up visits will be performed at 1, 2, 3, 6, 9, 12, and 24 months post system activation.
* A call visit will be performed at 18-months.
* All follow-up visits will require completion of a 3-day voiding diary by the patient before coming to the visit.
* During each clinic visit, stimulation parameters and level of treatment will be checked and adjusted as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Subject is at least 21 years old, with no plans to become pregnant during the trial. If of child bearing potential and sexually active, negative pregnancy test and using acceptable contraception.
3. Subject has been diagnosed with UUI for at least 6 months.
4. Subject experiences a minimum of four (4) leaking episodes associated with urgency, with at least one episode per day for 2 days documented on a voiding diary for 3 consecutive days.
5. If used, subject should be on stable dose of antimuscarinics and/or beta-3 adrenergic agonists for at least 1 month prior to baseline and agree to remain on stable medication consumption until the 24-month follow-up visit.
6. If used, subject should be on a stable dose of tricyclic antidepressants, Selective Serotonin Reuptake Inhibitors (SSRI) and Serotonin-Norepinephrine Reuptake Inhibitors (SNRI) for at least 3 months prior to baseline.
7. Subject agrees to attend all follow-up evaluations and is willing and capable to completely and accurately fill out voiding diaries and questionnaires and is willing to complete required exams and test

Exclusion Criteria:

1. Subject participation in a clinical investigation with an active treatment arm within the past 90 days.
2. Subject is a high surgical risk with multiple illnesses or active general infections that expose them to excessive bleeding or delayed or non-healing wounds. This includes patients who need anticoagulation therapy that cannot be temporarily stopped for the implantation procedure.
3. Subject with BMI >50.
4. Subject with any metal or other implant within 20cm distance of the area of BlueWind Revi implantation site.
5. Subject variation in diuretics consumption within the last 6 months.
6. Subject has received botulinum toxin injections for OAB within the past 12 months.
7. Subject with previous urinary incontinence surgery or prolapse surgery within the last 12 months.
8. Subject has had any spinal or genitourinary surgery within the last 6 months.
9. Subject had previous abdominoperineal resection of the rectum or radical hysterectomy (female)/ prostatectomy (male).
10. Subject with diagnosis of BPH with outflow/obstructive predominant symptoms.
11. Subject has skin, peripheral edema, orthopedic or neurologic anatomical limitations that preclude implantation or/and use of the device.
12. Subject with Alzheimer's, Parkinson, MS, stroke (CVI), neuropathy or injury resulting in neuropathy and/or suspected neurogenic bladder.
13. Subject has recurrent urinary tract infections (3 or more infections in the last 6 months), or presence of urinary fistula, or urinary tract obstruction such as cancer, urethral stricture or presence of urinary stone.
14. Subject with history of chemotherapy or pelvic radiotherapy that might have affected bladder control or caused neuropathies (i.e. peripheral neuropathy).
15. Male subject who have obstructive Benign Prostatic Hyperplasia (BPH) or other lower urinary tract obstructions.
16. Subject has open wounds or sores on the lower leg or foot or had previous, unhealed trauma in the implant area or has pitting edema (≥2+) in the lower leg.
17. Subject has Venous or Arterial disease/insufficiency in the lower leg or Vasculitis or dermatologic condition in the lower leg or infections near the implantation site in the lower leg.
18. Subject has a documented history of allergic response to Platinum iridium, Titanium, Zirconia, Gold, Silicone or Parylene.
19. Subject has other active implantable electronic device/s regardless of whether stimulation is ON or OFF.
20. Subject has a life expectancy of less than 1 year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | Month 4
  Superiority of active Revi therapy over non-active therapy in the treatment of subjects with urinary urge incontinence based on a 3-day voiding diary

CONTACTS AND LOCATIONS:
Overall Officials: Lori Fein, Study Director — BlueWind Medical
Locations (19):
- United States (19):
  - Arizona Urology Specialists, Tucson, Arizona
  - Pasadena Urology, Pasadena, California
  - Riverside Medical Clinic, Riverside, California
  - Florida Urology Partners, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Duly Health, Lombard, Illinois
  - Willis-Knighton Clinical Research, Shreveport, Louisiana
  - Chesapeake Urology, Owings Mills, Maryland
  - Specialty Clinical Research of St. Louis, LLC, St Louis, Missouri
  - Adult and Pediatric Urology and Urogynecology, Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - Duke Urogynecology - Duke University, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Sanford Female Pelvic Medicine & Reconstructive Surgery Clinic, Sioux Falls, South Dakota
  - Urology Partners of North Texas, Arlington, Texas
  - University of Texas Southwestern - Department of Urology, Dallas, Texas
  - DHR Health Institute for Research and Development, Edinburg, Texas
  - The Urology Place, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No